CLINICAL TRIAL: NCT00397527
Title: Safety Dermatological Evaluation: Acceptability With Gynecological Follow up of Dermacyd Wipes
Brief Title: Acceptability Dermacyd Wipes - Lactoserum - Hygiene
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LACTO_L_01810
Record Dates: First submitted 2006-11-08; First posted 2006-11-09 (Estimated); Last update posted 2008-05-16 (Estimated); Status verified 2008-05

CONDITIONS: Hygiene
MeSH Terms: interventions — lactoserum

INTERVENTIONS:
Drug: lactoserum

SUMMARY:
The purpose of this study is to demonstrate the safety of the gynecological formulation in normal and usual usage condition of Dermacyd Wipes

ELIGIBILITY:
The following information on clinical trials is provided for information purposes only to allow patients and physicians to have an initial discussion about the trial. This information is not intended to be complete information about the trial, to contain all considerations that may be relevant to potential participation in the trial, or to replace the advice of a personal physician or health professional.

Main criteria are listed hereafter:

Inclusion Criteria:

* Integral skin in the tested region

Exclusion Criteria:

* Pregnancy or breastfeeding women;
* Use of antiinflammatory or immunosuppression drugs;
* Topical medication use at the region to be treated;
* Cutaneous disease or active gynaecological disease which may interfer in study results;
* Personal history of allergic disease at the area to be treated;
* Allergic or atopic history.

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30
Dates: Start 2006-07

PRIMARY OUTCOMES:
Adverse events and their association with the treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Jaderson Lima, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis, São Paulo, Brazil